CLINICAL TRIAL: NCT02151162
Title: Mindfulness-Based Stress Management Program and Omega-3 Fatty Acids to Maintain Healthy Mental State in Hospital Nurses: Multi-Center Factorial-Design Randomized Controlled Trial Happy Nurse Project
Brief Title: Happy Nurse Project: Lifestyle Interventions to Maintain Healthy Mental State in Hospital Nurses
Acronym: HNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center of Neurology and Psychiatry, Japan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IRG-NP-NCNP-25-8
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Depressive Disorder; Anxiety Disorders
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Stress management plus omega-3 (Experimental): Thirty participants will be allocated to the arm. These interventions will terminate until 3 months from registration for each participant.
  Interventions: Behavioral: Mindfulness-based stress management program; Dietary Supplement: Omega-3 fatty acids pills
- Stress management plus placebo (Active Comparator): Thirty participants will be allocated to the arm. These interventions will terminate until 3 months from registration for each participant.
  Interventions: Behavioral: Mindfulness-based stress management program; Dietary Supplement: Placebo pills
- Psychoeducation leaflet plus omega-3 (Active Comparator): Thirty participants will be allocated to the arm. These interventions will terminate until 3 months from registration for each participant.
  Interventions: Dietary Supplement: Omega-3 fatty acids pills; Behavioral: Psychoeducation leaflet
- Psychoeducation leaflet plus placebo (Active Comparator): Thirty participants will be allocated to the arm. These interventions will terminate until 3 months from registration for each participant.
  Interventions: Behavioral: Psychoeducation leaflet; Dietary Supplement: Placebo pills

INTERVENTIONS:
Behavioral: Mindfulness-based stress management program — Mindfulness-based stress management program will be conducted by senior nurses in four individual sessions within these three months. Senior nurses have taken a 7-hour workshop including lectures and role-playing sessions. The detailed manual and videos including lectures will be provided to the senior nurses.
  Arms: Stress management plus omega-3; Stress management plus placebo
Dietary Supplement: Omega-3 fatty acids pills — Omega-3 fatty acids pills will include 1200 mg of eicosapentaenoic acid and 600 mg of docosahexaenoic acid per day.
  Arms: Psychoeducation leaflet plus omega-3; Stress management plus omega-3
Behavioral: Psychoeducation leaflet — Psychoeducation leaflet will include information about screening of stress, sleep hygiene, relaxation, and a list of consultants about mental health.
  Arms: Psychoeducation leaflet plus omega-3; Psychoeducation leaflet plus placebo
Dietary Supplement: Placebo pills — Placebo pills will include rapeseed oil, soybean oil, olive oil and fish oil.
  Arms: Psychoeducation leaflet plus placebo; Stress management plus placebo

SUMMARY:
The study is to explore the effectiveness of omega-3 fatty acids and mindfulness-based stress management program to maintain healthy mental state in hospital nurses. The participants will be junior nurses who work in inpatient wards and are not clinically depressed. The participants will be randomly allocated to four intervention arms: 1) Mindfulness-based stress management program plus omega-3 fatty acids pills ; 2) Mindfulness-based stress management program plus placebo pills; 3) Psychoeducation leaflet plus omega-3 fatty acids pills; and 4) Psychoeducation leaflet plus placebo pills. Thirty participants will be allocated to each arm. These interventions will terminate until three months from registration for each participant.

Information about depression and anxiety symptoms (primary outcome), insomnia, burnout, presenteeism, quality of life, sick leave, consultation about mental state of herself, and oxidative stress will be collected at 3 months, 6 months (primary time point) and 12 months from registration for each participant.

DETAILED DESCRIPTION:
The study is to explore the effectiveness of omega-3 fatty acids and mindfulness-based stress management program to maintain healthy mental state in hospital nurses. The participants will be junior nurses who work in inpatient wards at four general hospitals in Tama region in Tokyo, and are not clinically depressed based on the score of the Hospital Anxiety and Depression scale. The participants will be randomly allocated to four intervention arms: 1) Mindfulness-based stress management program plus omega-3 fatty acids pills; 2) Mindfulness-based stress management program plus placebo pills; 3) Psychoeducation leaflet plus omega-3 fatty acids pills; and 4) Psychoeducation leaflet plus placebo pills. Thirty participants will be allocated to each arm. These interventions will terminate until 3 months from registration for each participant. Stress management program will be conducted by senior nurses in four individual sessions within these three months. Psychoeducation leaflet will include information about screening of stress, sleep hygiene, relaxation, and a list of consultants about mental health.

Information about depression and anxiety symptoms (primary outcome), insomnia, burnout, presenteeism, quality of life, numbers of incident and accident at work, sick leave and consultation about mental state of herself, concentration of fatty acids in serum and oxidative stress will be collected at 3 months, 6 months (primary time point) and 12 months from registration for each participant. The primary outcome will be assessed by blind raters through telephone.

The outcomes will be compared between arms including stress management program and those without, and between arms including omega-3 fatty acids and those without, by using mixed model repeated measures model.

ELIGIBILITY:
Inclusion Criteria:

* Work for inpatient wards in among four general hospitals in Tama region, Japan, including: National Center of Neurology and Psychiatry Hospital, National Disaster Medical Center, Tokyo Metropolitan Tama Medical Center, and Tama-Hokubu Medical Center
* Nurses without administration work
* Give written consent in the participation of the study

Exclusion Criteria:

* Have plans to take sick leave, leave for other reasons or retirement within 26 weeks from the entry to the study
* Take structured psychotherapy (e.g. cognitive behavioral therapy, interpersonal therapy, and brief psychodynamic therapy) at the entry
* See a physician regularly in order to treat any mood or anxiety disorders primarily at the entry
* Take antidepressants, mood stabilizers, anticonvulsants or antipsychotics at the entry
* Have taken nutrient supplement including omega-3 fatty acids for 4 or more weeks within 52 weeks from the entry
* Clinically depressed, based on the total score of 11 or more on the Hospital Anxiety and Depression Scale - Depression Subscale and the total score of 15 or more on the Primary Health Care Questionnaire
* Consume 4 times or more of fish as the main course of meal per week
* Take anticoagulant drugs at the entry or have previous history of stroke or myocardial infarction
* Judged ineligible by research coordinator due to any reason

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-06-11 (Actual); Primary Completion 2016-03-02 (Actual); Study Completion 2016-09-06 (Actual)

PRIMARY OUTCOMES:
Blindly-rated depression and anxiety severity: Hospital Anxiety and Depression Scale (HADS) | 26 weeks
  The total score of the HADS (HADS-T) ranges from 0 to 42, with higher scores indicating more symptoms. The HADS has two sub scores, each ranging from 0 to 21: HADS-D (depression) and HADS-A (anxiety). The total score will be used as the severity of depression and anxiety symptoms in the present study.

SECONDARY OUTCOMES:
Blindly-rated depression and anxiety severity: Hospital Anxiety and Depression Scale (HADS) | 13 weeks
Blindly-rated depression and anxiety severity: Hospital Anxiety and Depression Scale (HADS) | 52 weeks
Major depressive episode: Primary Care Evaluation of Mental Disorders (PRIME-MD) | 26 weeks
  Major depressive episode will be ascertained using the Primary Care Evaluation of Mental Disorders (PRIME-MD) algorithm with the depression module of the Patient Health Questionnaire (PHQ-9). The PHQ-9 was developed as a self-report version of the PRIME-MD which aims at Diagnostic and Statistical Manual of Mental Disorders 4th edition (DSM-IV) diagnosis of several common mental disorders.
Major depressive episode: Primary Care Evaluation of Mental Disorders (PRIME-MD) | 13 weeks
Major depressive episode: Primary Care Evaluation of Mental Disorders (PRIME-MD) | 52 weeks
Depression severity: Personal Health Questionnaire-9 (PHQ-9) | 26 weeks
  Personal Health Questionnaire-9 is a 9-item structured questionnaire to measure depression severity.
Depression severity: Personal Health Questionnaire-9 (PHQ-9) | 13 weeks
Depression severity: Personal Health Questionnaire-9 (PHQ-9) | 52 weeks
Anxiety severity: Generalized Anxiety Disorder Assessment (GAD-7) | 26 weeks
  The GAD-7 consists of 7 items, and the total score ranges from 0 to 21.
Anxiety severity: Generalized Anxiety Disorder Assessment (GAD-7) | 13 weeks
Anxiety severity: Generalized Anxiety Disorder Assessment (GAD-7) | 52 weeks
Insomnia severity: Insomnia Severity Index (ISI) | 26 weeks
  The ISI is now considered a standard measure of the global severity of insomnia and used in many studies. The total score between 8-14 indicates subthreshold insomnia; and 15-28, clinical insomnia. The total score of the ISI will be used as the severity of insomnia in the study.
Insomnia severity: Insomnia Severity Index (ISI) | 13 weeks
Insomnia severity: Insomnia Severity Index (ISI) | 52 weeks
Somatic symptoms: The Bradford Somatic Inventory (BSI) | 26 weeks
  The BSI is a 44-item questionnaire for females about symptoms experienced in the previous month, which was designed to detect physical symptoms commonly related to depressed patients.
Somatic symptoms: The Bradford Somatic Inventory (BSI) | 13 weeks
Somatic symptoms: The Bradford Somatic Inventory (BSI) | 52 weeks
Presenteeism: World Health Organization Heath and Work Performance Questionnaire (HPQ) | 26 weeks
  The HPQ is a self-report instrument designed to estimate the workplace costs of health problems in terms of self-reported reduced job performance (presenteeism).
Presenteeism: World Health Organization Heath and Work Performance Questionnaire (HPQ) | 13 weeks
Presenteeism: World Health Organization Heath and Work Performance Questionnaire (HPQ) | 52 weeks
Burnout: Maslach Burnout Inventory (MBI) | 26 weeks
  The MBI is a self-report measure with 22 items and is calculated into three sub-domains such as emotional exhaustion, depersonalization and personal accomplishment.
Burnout: Maslach Burnout Inventory (MBI) | 13 weeks
Burnout: Maslach Burnout Inventory (MBI) | 52 weeks
Quality of Life: EuroQol (EQ-5D) | 26 weeks
  EQ-5D is a standardised instrument for use as a measure of health outcome. Applicable to a wide range of health conditions and treatments.
Quality of Life: EuroQol (EQ-5D) | 13 weeks
  EQ-5D is a standardised instrument for use as a measure of health outcome. Applicable to a wide range of health conditions and treatments.
Quality of Life: EuroQol (EQ-5D) | 52 weeks
  EQ-5D is a standardised instrument for use as a measure of health outcome. Applicable to a wide range of health conditions and treatments.

OTHER OUTCOMES:
Adverse events | 13 weeks
  Information about any possible adverse events will be collected during the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Norio Watanabe, MD, PhD, Principal Investigator — Kyoto University
Locations (2):
- Japan (2):
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
  - Kyoto University, Kyoto

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kunzler AM, Helmreich I, Chmitorz A, Konig J, Binder H, Wessa M, Lieb K. Psychological interventions to foster resilience in healthcare professionals. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD012527. doi: 10.1002/14651858.CD012527.pub2. PMID 32627860
- [Derived] Watanabe N, Horikoshi M, Shinmei I, Oe Y, Narisawa T, Kumachi M, Matsuoka Y, Hamazaki K, Furukawa TA. Brief mindfulness-based stress management program for a better mental state in working populations - Happy Nurse Project: A randomized controlled trial✰✰. J Affect Disord. 2019 May 15;251:186-194. doi: 10.1016/j.jad.2019.03.067. Epub 2019 Mar 22. PMID 30927579
- [Derived] Watanabe N, Furukawa TA, Horikoshi M, Katsuki F, Narisawa T, Kumachi M, Oe Y, Shinmei I, Noguchi H, Hamazaki K, Matsuoka Y. A mindfulness-based stress management program and treatment with omega-3 fatty acids to maintain a healthy mental state in hospital nurses (Happy Nurse Project): study protocol for a randomized controlled trial. Trials. 2015 Jan 31;16:36. doi: 10.1186/s13063-015-0554-z. PMID 25636180